CLINICAL TRIAL: NCT04564144
Title: A New Dual Function Oro-Dissolvable/Dispersible Meclizine HCL Tablet to Challenge Patient Inconvenience: In-Vitro Evaluation and In-Vivo Assessment in Human Volunteers
Brief Title: Evaluation of Meclizine Orodispersible Tablet Pharmacokinetic in Human Volunteers
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: meclizine pharmacokinetic
Record Dates: First submitted 2020-09-17; First posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Emesis
MeSH Terms: conditions — Vomiting | interventions — Meclizine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Volunteers receiving the prepared orodispersible tablets (Experimental): 6 human volunteers will receive the prepared orodispersible tablets plus a commercial one all containing Meclizine HCl in a parallel manner.
  Interventions: Drug: Meclizine Hydrochloride

INTERVENTIONS:
Drug: Meclizine Hydrochloride — A study will be conducted on the three tested orodispersible tablets and the commercial one (control). 6 volunteers are asked to cease any medication 7 days prior to blood sampling at least. Each volunteer will undergo 4 study sessions with one week of washout period in between (cross-overed to receive the other formulation). All volunteers are asked to fast overnight before taking the tablet. The tablet should be kept for 10 min in the mouth before swallowing without water. Just before taking the tablet, three milliliters of venous blood samples will be drown (predose, 0 h) and at 30, 60, 90, 120, 240, 360, 480, 720 min and 24 h postdose and stored in tubes coated with sodium heparin. Separation of plasma from Blood samples will be carried out by centrifuging at 5000 rpm for 10 min, then, it will be frozen at -20°C until analysis. By employing high-performance liquid chromatography (HPLC), the plasma concentration of MCZ will be assayed

SUMMARY:
The main goal of this study is to develop a new oro-dissolvable/dispersible tablet that will augment the dual rapid absorption of MCZ from the buccal cavity as well as prolonging that from the GIT. A dual function tablet is expected to encompass an outer coat of the drug with special excipients that will rapidly disperse and the drug get dissolve and absorb in the buccal cavity and an inner core that will similarly, disperse to release MCZ coated nanoparticles in the saliva. The latter will be subsequently swallowed without water to be absorbed in a prolonged manner from the GIT. This will be advantageous for geriatric as well as pediatric patients, besides, those suffering from dysphagia. The pharmacokinetics profile of the prepared dual function tablet will be assessed in human volunteers through noncompartmental analysis.

DETAILED DESCRIPTION:
The oral route is the most advantageous one for delivering drugs due to patient compliance and its convenient administration. Fast disintegrating drug delivery systems are those that disintegrate immediately in the buccal cavity liberating the drug which dissolves or disperses in the saliva without need of water. The European Pharmacopeia adopted oro-dispersible tablets (ODT) for a tablet that disintegrate or disperse in less than 60 sec in the buccal cavity before swallowing. So, the drug dissolution and absorption in addition to onset of clinical influence and drug bioavailability may be considerably better than those detected from conventional tablets and capsules. ODTs were initially industrialized to increase the patient compliance (children, geriatric and bedridden patients).

Nanoparticulate delivery systems have been investigated widely in the pharmaceutical industry owing to protection from degradation in GIT, the ability to control release of drugs and improvement of bioavailability.

Meclizine HCL, an antihistamine, has been widely used for prophylactic treatment of nausea, vomiting and management of dizziness accompanying motion sickness. MCZ is commonly used due to fewer adverse effects than other antihistaminic drugs but its onset of action is about 1 h and possesses short half-life. MCZ is a poor water soluble drug and associated with slow rate of absorption from oral route, therefore, there is a need to improve its dissolution and so ensure the maximum therapeutic utility. However, many different formulations of MCZ have been investigated to improve its overall solubility in order to enhance its bioavailability, such as; complexation with cyclodextrin, preparation of solid dispersions as oro- dispersible tablets and fast dissolving tablet by sublimation method. Moreover, authors will investigate the ability of floating microspheres to increase the half-life of MCZ

ELIGIBILITY:
Inclusion Criteria:

* Male aged between 30 and 40 years.
* Body weight range of 75kg-95kg.
* Healthy (defined as individuals who are free from significant nasal, cardiac, pulmonary, gastrointestinal, hepatic, renal, haematological, malignancy, endocrine, neurological and psychiatric disease as determined by history, physical examination and screening investigations).
* Non-smoking status. This can include ex-smokers who have given up smoking for >1 year.
* The subject is able and willing to give written informed consent to take part in the study and is available to complete all study measurements.

Exclusion Criteria:

* As a result of the medical interview, physical examination or screening investigations, the Investigator or appropriately qualified designee considers the subject unfit for the study.
* The subject has a history of drug or any other allergy, which, in the opinion of the Investigator or appropriately qualified designee, contraindicates their participation, including known or suspected personal history or family history of adverse reactions or hypersensitivity to anti histamines.
* The subject has participated in a study with a new molecular entity during the previous 3 months or any other study during the previous 2 months.
* The subject drinks alcohol.
* The subject is currently taking regular (or a course of) medication, prescribed (including all anti-allergy medication) or not (including over the counter medication or herbal remedies such as St Johns Wort). Paracetamol is an exception and will be permitted at daily doses of up to 4g following all doses of investigational product.
* The subject has tested positive for hepatitis C antibody or hepatitis B surface antigen.
* The subject has tested positive for HIV.
* The subject has a positive drugs of abuse and alcohol test.
* Donation of blood (450 mL or more) within 2 months of screening.
* Donation during the study would result in >500mL of blood being donated over a 56 day period
* Significant cardiac conduction abnormalities.
* Subjects with Perennial Allergic Rhinitis (PAR) and Seasonal Allergic Rhinitis (SAR), unless subjects with SAR are asymptomatic and it is outside of the pollen season
* Subjects who are unable to comply with study procedures.

Ages: 30 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — male
Enrollment: 6 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
measuring the Meclizine HCl plasma concentration | over 24 hours after dosing
  Using high performance liquid chromatography to measure the change in plasma drug concentrationز
measuring the Meclizine HCl Area under the curve | over 24 hours after dosing
  measuring the Meclizine HCl Area under the curve using high performance liquid chromatography
measuring the Meclizine HCl apparent clearance (CL/F) | over 24 hours after dosing
  measuring the Meclizine HCl apparent clearance (CL/F) using high performance liquid chromatography
measuring the maximum blood concentration of Meclizine HCl | over 24 hours after dosing
  measuring the maximum blood concentration of Meclizine HCl using high performance liquid chromatography
measuring the maximum blood concentration time of Meclizine HCl | over 24 hours after dosing
  measuring the maximum blood concentration time of Meclizine HCl using high performance liquid chromatography

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Y. Darwesh, Dr, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Dakhalia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang K, Li L, Song Y, Ye X, Fu S, Jiang J, Li S. Improvement of pharmacokinetics behavior of apocynin by nitrone derivatization: comparative pharmacokinetics of nitrone-apocynin and its parent apocynin in rats. PLoS One. 2013 Jul 30;8(7):e70189. doi: 10.1371/journal.pone.0070189. Print 2013. PMID 23936162
- [Result] Leach WT, Simpson DT, Val TN, Yu Z, Lim KT, Park EJ, Williams RO 3rd, Johnston KP. Encapsulation of protein nanoparticles into uniform-sized microspheres formed in a spinning oil film. AAPS PharmSciTech. 2005 Dec 6;6(4):E605-17. doi: 10.1208/pt060475. PMID 16408862
- [Result] Aljimaee YH, El-Helw AR, Ahmed OA, El-Say KM. Development and optimization of carvedilol orodispersible tablets: enhancement of pharmacokinetic parameters in rabbits. Drug Des Devel Ther. 2015 Mar 5;9:1379-92. doi: 10.2147/DDDT.S80294. eCollection 2015. PMID 25834396